CLINICAL TRIAL: NCT04849338
Title: The Role of Standardized Bleeding Score in Diagnosis of Pediatric Von Willebrand's Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Marina Kenz Basta, resident doctor at pediatric department sohag university hospital, Sohag University
Other Study IDs: Soh-Med-21-04-09
Record Dates: First submitted 2021-04-14; First posted 2021-04-19 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Von Willebrand's Diseased Children, Bleeding Questionnaire is Done

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Bleeding score ( questionnaire ) — Bleeding score is done for children diagnosed as von Willebrand's disease .

SUMMARY:
Von Willebrand's disease (VWD) is the most common inherited bleeding disorder. It arises from a deficiency in the quality or quantity of von Willebrand factor (VWF), a multimeric protein that is required for platelet adhesion. Typical patients present with mucocutaneous bleeding symptoms because of reduced circulating von Willebrand factor (VWF) In this study we will use the ISTH/SSC BLEEDING assessment tool as a standardized questionnaire and a proposal for a new bleeding score for inherited bleeding disorders

DETAILED DESCRIPTION:
Von Willebrand's disease (VWD) is the most common inherited bleeding disorder. It arises from a deficiency in the quality or quantity of von Willebrand factor (VWF), a multimeric protein that is required for platelet adhesion. Typical patients present with mucocutaneous bleeding symptoms because of reduced circulating von Willebrand factor (VWF) . A predictive bleeding score could reveal individuals who may benefit from repetitive testing and those for whom repetitive testing is unlikely to be of benefit . In 2005, Rodeghiero, et al. developed a standardized questionnaire for the evaluation of haemorrhagic symptoms, referred to hereafter as the Vicenza score. Their retrospective analysis found that >3 haemorrhagic symptoms or bleeding scores of 3 in men and 5 in women was very specific (98.6%) for VWD, although less sensitive (69.1%)]. These investigators later reported in a larger population that higher bleeding scores were associated with increasing likelihood of VWD and bleeding after surgery or tooth extraction. Neither of these studies prospectively surveyed paediatric populations. As a result of their shorter life experience, children have fewer exposures to bleeding challenges such as dental extractions, surgeries, menarche and childbirth. In 2009, Bowman, et al. administered a modified Vicenza bleeding score to a naive primary care paediatric population and determined a bleeding score ≥2 was abnormal. Using this definition, their bleeding score had a high negative predictive value (0.99) and could accurately distinguish between children with and without VWD. In this study we will use the ISTH/SSC BLEEDING assessment tool as a standardized questionnaire and a proposal for a new bleeding score for inherited bleeding disorders. For each specific bleeding symptom, the ISTH/SSC joint working group proposed minimal criteria in order to classify a symptom as significant and thus receive a score of 1 or more. Symptoms included in this questionnaire are epistaxis , cutaneous bleeding , minor cutaneous wound , oral cavity bleeding , hematemesis , melena and hematochezia , hematuria , tooth extraction , surgical bleeding , menorrhagia , postpartum bleeding , muscle hematomas or hemoarthrosis and CNS bleeding .

ELIGIBILITY:
Inclusion Criteria:

* This study included children, aged 1 week-18 years, referred to Sohag university hospital for evaluation of bleeding symptoms, family history of a bleeding disorder and/or abnormal coagulation studies.
* Bleeding questionnaire is done during patients' clinic visit.

Exclusion Criteria:

1. Patients older than 18 years.
2. Other inherited or acquired bleeding disorders.
3. Patients on regular antiplatelets or anticoagulants.

Inclusion Criteria:

* This study included children, aged 1 week-18 years, referred to Sohag university hospital for evaluation of bleeding symptoms, family history of a bleeding disorder and/or abnormal coagulation studies.
* Bleeding questionnaire is done during patients' clinic visit.

Exclusion Criteria:

1. Patients older than 18 years.
2. Other inherited or acquired bleeding disorders.
3. Patients on regular antiplatelets or anticoagulants.

Ages: 1 Week to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: children, aged 1 week-18 years, referred to Sohag university hospital , von Willebrand's diseased
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-04-15 (Estimated); Primary Completion 2022-05-15 (Estimated); Study Completion 2022-05-15 (Estimated)

PRIMARY OUTCOMES:
Use bleeding score as diagnostic tool of von Willebrand's disease | Within one year
  The aim of the present study is to assess the diagnostic power of the bleeding score in identifying VWD in a prospective cohort of patients referred to a paediatric haematology clinic for evaluation of a bleeding disorder , so we can predict the next bleeding episode and minimize the complications

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol